CLINICAL TRIAL: NCT05156372
Title: Pilot Study of a Randomized Chemo-periodized Adjuvant High-Intensity Interval Training Intervention to Improve Chemotherapy Tolerance in Men With Metastatic Prostate Cancer
Brief Title: Adjuvant High-intensity Interval Training During Chemotherapy in Metastatic Prostate Cancer Patients
Acronym: HIIT PCa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution, no subjects were enrolled
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTMS 21-0078; HSC20210663H (Other: UT Health San Antonio)
Record Dates: First submitted 2021-09-29; First posted 2021-12-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer Metastatic; Castrate Resistant Prostate Cancer; Metastatic Prostate Cancer; Metastatic Prostate Adenocarcinoma
Keywords: metastatic prostate cancer; high-intensity interval training; HIIT; exercise; exercise oncology; resistance training
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessments and analysis will be done by study staff blinded to the participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants will engage in 2-3 supervised high intensity aerobic and resistance exercise sessions per week.
  Interventions: Other: High Intensity Interval Training
- Control (No Intervention): Participants will continue daily routine as usual and given an informational flyer on physical activity and cancer.

INTERVENTIONS:
Other: High Intensity Interval Training — Participants will perform high-intensity aerobic and resistance exercise
  Other Names: HIIT
  Arms: Exercise Intervention

SUMMARY:
This study aims to examine the use of high-intensity interval training (HIIT) and resistance training on docetaxel chemotherapy tolerability and toxicity in metastatic prostate cancer.

DETAILED DESCRIPTION:
Exercise has been shown to decrease tumor progression and mitigate treatment-related side effects, such as fatigue, while increasing physical fitness. In this study, investigators will test the effects of a high intensity interval training and resistance exercise program on how patients with metastatic prostate cancer tolerate docetaxel chemotherapy. Participants assigned to the exercise intervention will be asked to meet with a personal trainer 2-3 times per week for supervised exercise sessions. All participants will be asked to complete electronic questionnaires during their chemotherapy sessions that ask about their physical and mental wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic prostate cancer

  * Includes metastatic hormone sensitive prostate cancer, AND
  * Metastatic castration resistant prostate cancer
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Planned to receive docetaxel chemotherapy for treatment of prostate cancer with plan for at least 4 cycles of therapy
* Estimated life expectancy > 6 months
* Must be receiving androgen deprivation therapy (ADT) during study period or have had prior bilateral orchiectomy
* 4 weeks from any major surgery
* Age > 18 years
* Willing to participate in exercise intervention per protocol
* Cleared by study personnel to participate in exercise intervention based on screening physical exam
* Eligible patients can be participating in other investigational protocols or consent to other investigational protocols during this study participation if it does not affect docetaxel dosing, include additional cytotoxic chemotherapy, or interfere with exercise intervention
* Patients must be able to travel to one of the study-designated exercise facilities up to three days per week
* Required Initial Laboratory Values:

  * Absolute neutrophil count (12) ≥ 1500/uL
  * Platelet count ≥ 100,000/uL
  * Creatinine ≤ 1.5 x upper limits of normal
  * Bilirubin ≤ 1.5 x upper limits of normal
  * Aspartate aminotransferase (AST) ≤ 1.5 x upper limits of normal
  * Serum testosterone ≤ 50 ng/dL

Exclusion Criteria:

* Known small cell neuroendocrine cancer of the prostate
* Has already initiated first-line chemotherapy treatment course
* Poorly controlled hypertension, BP >160/90 on >1 occasion during screening period
* NYHA Class II heart failure
* Serious cardiovascular event within 6 months of consent, including transient ischemic attack, cerebrovascular accident, or myocardial infarction
* Receiving additional cytotoxic chemotherapy in addition to docetaxel during study participation
* Stable or unstable angina
* Active second malignancy, with exception of non-melanoma skin cancer or non-invasive bladder cancer
* Known physical limitation that would impede participation in exercise per protocol
* Moderate-to-severe bone pain (i.e NCI common terminology criteria of adverse events grade 2-3 bone pain)
* Men already participating in vigorous aerobic exercise for more than 60 minutes per day or structured resistance exercise (>2 upper body and >2 lower body exercises) 2 or more days a week.
* Psychiatric illness, which would prevent the patient from giving informed consent or adhering to the study protocol.
* Has chest pain during physical activity (patient can participate with cardiologist clearance).
* Uncontrolled asthma (patient can participate if on asthma controlling medications and has access to rescue inhaler).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Docetaxel chemotherapy tolerability | 2 years
  Number of Changes or delays in docetaxel treatment schedule or dosing (tolerability)
Docetaxel chemotherapy toxicity | 2 years
  Rates of CT CAE v.5 reported symptoms related to treatment
Functional assessment of Cancer therapy (FACT)-Taxane subscale | Baseline to 2 years
  Change in score on a 16 point scale using a 5-point response scale focused on patient-reported neuropathic symptoms and concerns:
  0 =Not at all
  1. =A little bit
  2. =Somewhat
  3. =Quite a bit
  4. =Very much
  Range of scores is from 0-64 with a lower score indicating less neuropathic symptoms and concerns.

SECONDARY OUTCOMES:
Functional assessment of Cancer therapy (FACT)-G | Baseline to 2 years
  Change in FACIT-G score. FACT-G contains four subscales measuring physical well being, social well-being, emotional well-being, and functional well being containing 7,7,6, and 7 items respectively. Responses to questions are scored:
  0 =Not at all
  1. =A little bit
  2. =Somewhat
  3. =Quite a bit
  4. =Very much
  Scores from the 4 scales are added to give a total score between 0-108, where a lower score indicates better physical, social, emotional and functional well-being.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline to 2 years
  Change in score on this subscale, which contains 13 items assessing the consequences of fatigue. Each item is rated on a 5-point Likert scale ranging from 0=not at all to 4=very much.
  Totals range from 0-52 with a lower score indicating less fatigue.
European Organization for Research Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline to 2 years
  Change in score for 30 questions to assess the quality of life with 9 multi-item scales: 5 functional scales; 3 symptom scales; and a global health and quality-of-life (GHQL) scale. A few 1-item symptom measures are included. Score is calculated from the mean of 13 of the 15 QLQ-C30 scales (GHQL and the Financial Impact scale are not included). Prior to calculating the mean, the symptom scales are reversed to obtain a uniform direction of all scales.
  All scales and 1-item measures range from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Pittsburgh Sleep Quality Index (PSQI) | Baseline to 2 years
  Change in score on this 19-question assessment will be used to assess sleep quality and sleep habits.
  The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Godin Leisure | Baseline to 2 years
  Change in score calculated using the following formula: Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light). The first 3 questions relate to type of activity and the 4th to number of times a week the activity is engaged in for at least 15 minutes.
  EXAMPLE Strenuous = 3 times/wk Moderate = 6 times/wk Light = 14 times/wk Total leisure activity score = (9 × 3) + (5 × 6) + (3 × 14) = 27 + 30 + 42 = 99
  Godin Scale Score: Interpretation 24 units or more: Active 14-23 units: Moderately Active Less than 14 units: Insufficiently Active/Sedentary

OTHER OUTCOMES:
Serum inflammatory biomarkers associated with tumor progression | 2 years
  Compare changes in levels of serum measurements of biomarkers such as tumor necrosis factor alpha (pg/ml) and interleukins (pg/ml).
Body Composition | 2 years
  Compare changes in fat free mass and fat mass measured with dual energy x-ray absorptiometry (DEXA) scan from baseline to end-of-study
Muscular Strength | 2 years
  Compare changes in participant's 1 repetition maximum (1RM) weight between baseline and end-of-study for chest press, leg press, seated row, leg extension, and grip strength. Participants will lift progressively heavier weight in each exercise until unable to lift any extra weight. This will be recorded as the 1RM weight. Total load will be calculated across exercises, with higher load values indicating higher muscular strength.
Aerobic Fitness | 2 years
  Compare participant's time to completion on a 400 meter walk test from baseline to end-of-study. This submaximal test serves as a surrogate measure of aerobic fitness.
Cognitive function changes over time | 2 years
  Compare cognitive function changes between groups over time measured by Cambridge Neuropsychological Test Automated Battery (CANTAB).

CONTACTS AND LOCATIONS:
Overall Officials: Darpan I Patel, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No